CLINICAL TRIAL: NCT00995956
Title: Quantitative Measurements of Albumin, Total and Free Fraction of Mycophenolic Acid, and Measurement of IMPDH Activity in Liver Transplants.
Brief Title: Albumin, Total and Free Fraction of Mycophenolic Acid, and Measurement of IMPDH Activity in Liver Transplants.
Acronym: Albumix
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Pål Aarstrand Reine, Mr, Oslo University Hospital
Other Study IDs: 2009/716a
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Liver Transplant
Keywords: Albumin; Mycophenolic acid; IMPDH; Free fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for drug analyzes
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study we aim to investigate to what extent the serum albumin concentration in liver transplant patients treated with mycophenolic acid (MPA) affect the free fraction of MPA. Furthermore we will investigate if a change in free fraction has implications for the immunosuppressive effect of MPA by measuring the IMPDH activity. This might in the future provide opportunity for further individualisation of the treatment with MPA. We will also investigate if the stabilizers present in pharmaceutical-grade albumin have a displacement effect on MPA in Vitro (ref).

DETAILED DESCRIPTION:
This is a prospective, open, non randomised study without intervention. Our main goal is to find out what effect the albumin concentration has on the free fraction MPA and IMPDH activity in the lymphocytes.

There will be taken blood samples on day 2, 3 or 4 after transplantation. There will be taken one sample before intake of MPA then another 8 samples during the next 4 hours. The samples will be analyzed with regards to MPA and IMPDH. We will follow the progress of free fraction MPA and IMPDH activity (variables; area under the curve, maximum value, minimum value, time to max and min)

The results will be correlated with the other laboratory results and clinical data. In addition to our main aim, to find correlation between free fraction MPA and albumin values, we will describe the relationship between free fraction MPA and IMPDH activity. We will also study the effect on free fraction MPA after adding stabilizers present in pharmaceutical-grade albumin to our serum samples.

The samples will be taken from an indwelling central venous catheter routinely introduced during the transplant surgery. The drug analyses will be performed by the Section for analytic pharmacology and endocrinology. MPA concentrations will be measured by a method based on HPLC with UV-detection. Enzymatic activity for IMPDH will be analysed by a validated method developed in-house (ref). Other biochemical analyzes included in this study is routinely analyzed in liver transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant, MPA treatment

Exclusion Criteria:

* malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant pations from Rikshospitalet HF
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf E Kongsgaard, Prof, Study Chair — Oslo University Hospital
Locations (1):
- Oslo university Hospital, Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Reine PA, Kongsgaard UE, Andersen A, Thogersen AK, Olsen H. Infusion of albumin attenuates changes in serum protein binding of drugs in surgical patients compared with volume replacement with HAES. Acta Anaesthesiol Scand. 2008 Mar;52(3):406-12. doi: 10.1111/j.1399-6576.2007.01555.x. PMID 18269390
- [Background] Vethe NT, Bergan S. Determination of inosine monophosphate dehydrogenase activity in human CD4+ cells isolated from whole blood during mycophenolic acid therapy. Ther Drug Monit. 2006 Oct;28(5):608-13. doi: 10.1097/01.ftd.0000245680.38143.ca. PMID 17038874